CLINICAL TRIAL: NCT02516761
Title: Effect of Low-impact Aerobic Exercise Combined With Music Therapy in Patients With Fibromyalgia
Brief Title: Effect of Low-impact Aerobic Exercise and Music Therapy in Fibromyalgia
Acronym: EffMusFibro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Ph, D, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ID011
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Music Therapy; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-impact aerobic exercise combined with music therapy (Experimental): Intervention consists in working the muscles which are mostly affected by fibromyalgia through group exercises, which are dynamic, smooth and aim functionality. This exercise is done to the rhythm of melodic music, adapted to the tastes of the participants and also adapted on the way to perform the exercise.
  Interventions: Other: Low-impact aerobic exercise combined with music therapy
- Low-impact aerobic exercise (Experimental): Then intervention is like the previous group but with the difference that physical activity is not performed to the rhythm of chosen melodic music. Therefore, exercises are done with general chill-out music throughout the session, without adaptation of the exercise to the music.
  Interventions: Other: Low-impact aerobic exercise
- Control group (Active Comparator): With this group no intervention is done, but they are assessed like the other groups.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Low-impact aerobic exercise combined with music therapy — Intervention consists in working the muscles which are mostly affected by fibromyalgia through group exercises, which are dynamic, smooth and aim functionality. Each session consists of 60 minutes with 3 parts: initial warming up time, main part through games, group dynamics and pure aerobic workout, and final cool down with stretching. This exercise is done to the rhythm of melodic music, adapted to the tastes of the participants and also adapted on the way to perform the exercise. For this, they were shown a list of 100 music compositions from which participants choose a minimum of 20 preferences. All exercises are performed with proper postural control both dissociated and global and within a framework of therapeutic proprioceptive gymnastics.
  Arms: Low-impact aerobic exercise combined with music therapy
Other: Low-impact aerobic exercise — Low-impact aerobic exercise. Then intervention is like the previous group but with the difference that physical activity is not performed to the rhythm of chosen melodic music. Therefore, exercises are done with general chill-out music throughout the session, without adaptation of the exercise to the music.
  Arms: Low-impact aerobic exercise
Other: Control group — With this group no intervention is done, but they are assessed like the other groups.
  Arms: Control group

SUMMARY:
The idea of this study is the combination of these two techniques (low-impact aerobic exercise through functional movements and music therapy) that have proven to be effective separately. The main objective of this study is to test this combination to reduce widespread pain in fibromyalgia patients, improve their balance, influence on decreasing levels of depression and improve quality of life.

DETAILED DESCRIPTION:
Material and methods Patients The sample includes volunteer subjects diagnosed with fibromyalgia from the Valencian Association of People Affected by Fibromyalgia that were submitted to participate in the study.

Study design It is a quasi-experimental, longitudinal, prospective, controlled, randomized, single-blinded research. The sample was divided into 3 groups. Patients signed informed consent and then the randomization of subjects to the different study groups was done through computer software by an external assistant who was blinded to the study objectives. The study was conducted in morning and afternoon sessions.

All those patients who belong to the experimental group 1 or 2 attend their sessions which last 60 minutes and are held 2 times a week every other day. The experimental group 1 attends classes in the morning, while the experimental group 2 attends them in the evenings. The control group only comes to the evaluation sessions without doing any particular activity. The subjects are evaluated in two stages, at baseline and after completion of the study.

Intervention Group 1 (G1): Low-impact aerobic exercise combined with music therapy. Intervention consists in working the muscles which are mostly affected by fibromyalgia through group exercises, which are dynamic, smooth and aim functionality.

Group 2 (G2): Low-impact aerobic exercise. Then intervention is like the previous group but with the difference that physical activity is not performed to the rhythm of chosen melodic music. Therefore, exercises are done with general chill-out music throughout the session, without adaptation of the exercise to the music.

Control group (CG): With this group no intervention is done, but they are assessed like the other groups.

Evaluation:

Depression, by Beck Depression Inventory, General discomfort, using the Faces Pain Scale, Balance, evaluated by the Berg Scale.

ELIGIBILITY:
Inclusion Criteria:

* To be between 30 and 80 years old.
* Meet the new diagnostic criteria for fibromyalgia of the ACR..
* Meet some or several of the following characteristics:

  * Depression
  * Anxiety
  * Muscle pain
  * Fatigue
  * Sleep disturbance
* May have limited mobility as long as it is caused by fibromyalgia.

Exclusion Criteria:

* Medical contraindication for physical activity (locomotor disorder, uncontrolled cardiovascular disease, ...)
* Deafness or limited hearing
* Vestibular disorders that compromise balance.
* Very low visibility or blind people.
* Psychiatric disorders or excessive emotional tension that could alter the dynamics of the study (psychotic disorder)
* Cognitive disabilities
* Decompensation or changes in medication.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
General discomfort. | 8 weeks
  General discomfort, using the Faces Pain Scale. This scale assesses in a global way widespread pain of patients. It values from 0 to 10 on a scale of facial expression (0 = no pain and smiling face, up to 10 = worst possible pain and sad face). The reliability coefficient for this scale is Cohen = 0.61.

SECONDARY OUTCOMES:
Depression. | 8 weeks
  By Beck Depression Inventory. This scale aims to assess depression and its somatic intensity by 21 different items assessing depressive symptoms. It includes four answer options arranged from lowest to highest severity. This version is adapted to Spanish and validated and has an internal consistency with Cronbach's alpha coefficient = 0.83. The scale emphasizes more on the cognitive component of depression (15 items), being the symptoms of somatic / vegetative type the second most important group (6 items). The result of 0-9 points means that there is no depression, 10 to 18 points mild depression, 19-29 moderate depression and 30 points indicates severe depression.
Impact on quality of life. | 8 weeks
  The Fibromyalgia Impact Questionnaire (FIQ).It is a multidimensional self-administered questionnaire with 10 items that evaluates the status of the patient the week before the test is filled, and it assesses the aspects that tend to be more affected in people with fibromyalgia. The first item contains 10 sub-items, ranging from 4 points (from = always to 3 = never) and assesses the patient's functional capacity in activities of daily living. The second and third item refers to days of the week and the rest are visual analog scales from 0 to 10. This scale was validated in its Spanish version in 2013, obtaining a Cronbach coefficient= 0.95.
Balance. | 8 weeks
  Evaluated by the Berg Scale. Scale on which the balance is evaluated and consists of 14 items, which assess the change of position from sitting to standing position, as well as standing and sitting position without assistance, transfers, standing with eyes closed, feet together, one foot advanced, one leg support, inclination of the body, the ability to pick up an object from the floor and also to turn around (to look back only, or giving a full turn). The internal consistency of the questionnaire is alpha 0.98 and test-retest reliability of 0.98 with a range of 0.86 to 0.99 for individual items.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V gemma.espi@uv.es, P, Study Director — Department of Physiotherapy
Locations (1):
- Gemma V. Espí López, Valencia, Valencia, Spain

REFERENCES:
- [Result] Wolfe F, Walitt BT, Rasker JJ, Katz RS, Hauser W. The Use of Polysymptomatic Distress Categories in the Evaluation of Fibromyalgia (FM) and FM Severity. J Rheumatol. 2015 Aug;42(8):1494-501. doi: 10.3899/jrheum.141519. Epub 2015 Jun 15. PMID 26077414
- [Result] Kajantie E, Phillips DI. The effects of sex and hormonal status on the physiological response to acute psychosocial stress. Psychoneuroendocrinology. 2006 Feb;31(2):151-78. doi: 10.1016/j.psyneuen.2005.07.002. Epub 2005 Sep 1. PMID 16139959
- [Result] de Miquel CA, Campayo J, Florez MT, Arguelles JM, Tarrio EB, Montoya MG, Martin A, Salio AM, Fuentes JV, Alberch EA, de la Camara AG. Interdisciplinary consensus document for the treatment of fibromyalgia. Actas Esp Psiquiatr. 2010 Mar-Apr;38(2):108-20. PMID 21361054